CLINICAL TRIAL: NCT07186335
Title: Effectiveness of Promoting the Role of General Practitioners in a Mental Health Care System Integrated With Primary Care in Adolescence, According to the World Health Organization Definition
Acronym: MGIntegrADO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Santé des Étudiants de France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00883-42
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Adolescent Behavior
Keywords: teenagers and young adults; general practitioner
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: self-questionnaire — Quantitative survey with self-administered questionnaire offered to all patients

SUMMARY:
MG-integr-ADO aims to create and evaluate in France, a system of integrated mental health care in primary care for adolescents with mental illness.

The objective is to show that an intervention promoting the role of the general practitioner in the continuity of mental health care for young people with a team of "Indicated primary preventive interventions" (Relay) increases the rate of patients for whom the general practitioner has been contacted (presence of at least one contact with the general practitioner of the adolescent whether by telephone, mail or email, traced in the file) between the beginning and the end of care

DETAILED DESCRIPTION:
Non-interventional multicenter prospective mixed study

Research process in 3 phases:

1. multi-method inventory :

   a : Systematic review of the international literature on integrated mental health systems in primary care (done), b : Quantitative component evaluating the effective number of contacts of the general practitioner (front) in the Relays, c : Qualitative section on the Relay-general practitioner link (Interviews with Relay Professionals, GPs, patients)
2. construction and deployment of the intervention to create the integrated system
3. after the intervention, evaluation of its effect (number of general practitioners contacted, evolution at 6 months of adolescents treated: somatic and psychic state, unscheduled care, satisfaction)

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 11-25 suffering from mental health issues
* Living in the relevant health region
* Attending Relais d'Ile-de-France centers (75, 77, 92, 93) alone or accompanied by someone

Exclusion Criteria:

* Young people outside the 11-25 age group - Parents and children who do not speak French or cannot read or write.
* Refusal to participate
* Young people in crisis situations requiring immediate hospitalization without care at Le Relais.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Young people aged 11-25 who have consulted the FSEF's Relais services, parents of these young people, Relais professionals, general practitioners
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
comparaison | self-questionnaire
  The percentage of young people for whom the general practitioner was contacted between the start (known as T0) and the end of care (known as T1), as reported by the young person.
  [Time Frame: To the inclusion of young people and in the End of care (care between 6 months to 1 year)]

IPD SHARING:
Plan to Share IPD: No